CLINICAL TRIAL: NCT06413225
Title: Multi-centre Post-Market Data Collection Protocol to Evaluate the Performance of Synergy Spine Solutions Synergy Disc®
Brief Title: Multi-Centre Post-Market Data Collection
Status: Withdrawn | Type: Observational
Why Stopped: Multiple sites in the UK, went to EC for multicenter approval after this record was written
Sponsor: Synergy Spine Solutions (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 21-001-UK01
Record Dates: First submitted 2024-04-22; First posted 2024-05-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: radiculopathy; myelopathy; disc replacement; motion preservation
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: All patients for whom the decision has been made to have the Synergy Disc system implanted and give informed consent will be enrolled in this study, following country-specific requirements.
  Interventions: Device: Synergy cervical disc system
- Retrospective: Patients who have previously received the Synergy Disc system in the last ten years are eligible for inclusion in the retrospective data collection; a waiver of consent, or an informed consent, for the retrospective data collection from the medical records of the implanting surgeon will be sought per country-specific regulations.
  Interventions: Device: Synergy cervical disc system

INTERVENTIONS:
Device: Synergy cervical disc system — motion preservation disc

SUMMARY:
This is a real world data collection observational study at a single site. There are both prospective and retrospective cohorts. The study will examine the safety and effectiveness of the Synergy cervical disc system in patients with degenerative cervical disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 or above at the time of the surgery.
2. Have had (retrospective cohort) or the decision has been made to have (prospective cohort) the Synergy Disc implanted
3. Skeletally mature patients for reconstruction of the disc from C3-C7 following a single or multiple level discectomy for intractable radiculopathy
4. Intractable radiculopathy and/or myelopathy with at least one of the following producing symptomatic nerve root and/or spinal cord compression:

   1. herniated disc and/or osteophyte formation
   2. Symptomatic nerve root and/or spinal cord compression documented by patient history (arm or neck pain and/or neurologic deficit) and imaging (CT, MRI, x-rays, etc.)
   3. Failed a minimum of 6 weeks conservative treatment
5. Written informed consent given by subject

Exclusion Criteria:

* Inclusion Criteria: All answers must be YES to be eligible for the study.

  1. Age 21 or above at the time of the surgery.
  2. Have had (retrospective cohort) or the decision has been made to have (prospective cohort) the Synergy Disc implanted
  3. Skeletally mature patients for reconstruction of the disc from C3-C7 following a single or multiple level discectomy for intractable radiculopathy
  4. Intractable radiculopathy and/or myelopathy with at least one of the following producing symptomatic nerve root and/or spinal cord compression:

     1. herniated disc and/or osteophyte formation
     2. Symptomatic nerve root and/or spinal cord compression documented by patient history (arm or neck pain and/or neurologic deficit) and imaging (CT, MRI, x-rays, etc.)
     3. Failed a minimum of 6 weeks conservative treatment
  5. Written informed consent given by subject

Exclusion Criteria: All answers must be NO to be eligible for the study.

1. Moderate to advanced spondylosis
2. Diagnosis of osteoporosis
3. Active systemic infection or infection at the operative site
4. Pregnancy
5. Marked cervical instability on lateral, coronal, or flexion/extension radiographs
6. Cervical spine condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level
7. Severe pathology of the facet joints of the involved vertebral bodies
8. Previous diagnosis of osteopenia or osteomalacia
9. More than one immobile vertebral level between C1 and T1 from any cause
10. Morbid obesity
11. Vulnerable person (pregnant patients, emergency cases, children, prisoners and people without mental capacity)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People over the age of 21 diagnosed with cervical degenerative disc disease and for whom the Synergy Disc device is an option (prospective cohort) or has already been implanted (retrospective cohort).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2029-09-25 (Estimated); Study Completion 2034-09-25 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 12 months
  Neck disability Index improvement of >15 pts (out of 100) in subjects by 12 months post operative compared with baseline. A lower score is a better score.
device Related or Device Procedure Related Adverse Events | 12 months
  Absence of major device related adverse events defined as radiographic failure, neurologic failure or failure by adverse event

SECONDARY OUTCOMES:
Visual Analog Scale Neck and Arm Pain Measurement | pre-operative, 6 week, 3 month, 6 month, 12 month, annually post-operatively
  Pain will evaluated by the Visual analog scale (VAS) (place a line from zero where there is no pain to 10 which is the worst pain imaginable), by NRS (circle a number from zero to ten where zero equals no pain and ten is worst imaginable) to or a verbal description that the doctor writes down, per the site's Standard of Care. A change of at least 20 mm will be considered clinically significant. Neck pain as measured on a 100mm VAS at baseline and at each follow-up timepoint. Left and Right arm/shoulder pain as measured on a 100 mm VAS at baseline and at each follow up time-point.
Patient Satisfaction | 6 week, 3 month, 6 month, 12 month, annually post-operatively
  patient completed questionnaire on their satisfaction with the disc replacement surgery
Motor and Sensory Function in the Arm | pre-operative, 6 week, 3 month, 6 month, 12 month, annually post-operatively
  maintenance or improvement in neurologic status compared with baseline will be assessed using a defined numeric scale ranging from 0 (normal) to 5 (deficit)
Nurick's Criteria | pre-operative, 6 week, 3 month, 6 month, 12 month, annually post-operatively
  Disease status as characterized by physician at each time point
Odom's criteria | 6 week, 3 month, 6 month, 12 month, annually post-operatively
  surgical outcome characterized by physician at each post operative visit

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Orthopedic Hospital, Birmingham
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No